CLINICAL TRIAL: NCT05718037
Title: A Phase I, Randomized, Observer-blinded Study to Evaluate the Safety, Tolerability, and Immunogenicity of BV211 in Adult Volunteers
Brief Title: Phase I Clinical Trial of a Candidate Herpes Zoster Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan BravoVax Co., Ltd. (Industry)
Collaborators: Shanghai BravoBio Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BV-C211-202301
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster Vaccine; BV211
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LY (Experimental): Young adult subjects received low dose of BV211
  Interventions: Biological: Recombinant Zoster Vaccine
- HY (Experimental): Young adult subjects received high dose of BV211
  Interventions: Biological: Recombinant Zoster Vaccine
- Placebo (Placebo Comparator): Young adult subjects received placebo
  Interventions: Biological: Placebo
- LO (Experimental): Old adult subjects received low dose of BV211
  Interventions: Biological: Recombinant Zoster Vaccine
- HO (Experimental): Old adult subjects received high dose of BV211
  Interventions: Biological: Recombinant Zoster Vaccine
- Control Vaccine (Active Comparator): Old adult subjects received control vaccine
  Interventions: Biological: Zoster Vaccine Recombinant, Adjuvanted

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine — 0.5mL, Intramuscular
  Other Names: BV211
  Arms: HO; HY; LO; LY
Biological: Placebo — 0.5mL, Intramuscular
  Arms: Placebo
Biological: Zoster Vaccine Recombinant, Adjuvanted — 0.5mL, Intramuscular
  Other Names: Shingrix
  Arms: Control Vaccine

SUMMARY:
This is a phase I, randomized, observer-blinded study to evaluate the safety, tolerability, and immunogenicity of BV211(a herpes zoster vaccine) in Adult Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy resident aged 30-70 years with body weight ≥ 50 kg for males and ≥ 45 kg for females, BMI within the range of 19.0-32.0 (including the boundary value), who can provide legal identification.
* Willing to participate in the study and sign ICF.
* Women of childbearing age shall take effective contraception measures 30 days before vaccination up to 6 months post full vaccination and not in lactation period. The pregnancy test on the day of vaccination shall be negative.
* Will attend all scheduled follow-up visits and follow the requirements of the clinical study.

Exclusion Criteria:

* Smoking, and/or excessive alcohol use.
* Failed the screening test of illicit drugs, including THC.
* Axillary temperature above 37.3℃.
* History of herpes zoster.
* Received any herpes zoster vaccine.
* Received any vaccine within 14 days or live vaccine within 28 days before vaccination.
* Received gamma immunoglobulin or intravenous immunoglobulin within 3 months before vaccination.
* Have acute illness or are in the acute exacerbation phase of a chronic disease within 3 days before vaccination.
* Allergic history to any vaccine-related component; history of severe allergies to any vaccine.
* History of convulsions, epilepsy or encephalopathy (such as congenital brain hypoplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral infarction, brain infection, damage to nerve tissue in brain caused by chemical drug poisoning, etc.) and psychiatric history or family history of mental illness.
* Asplenia or functional asplenia, and asplenia or splenectomy caused by any reason.
* Primary or secondary immunocompromised or diagnosed with congenital or acquired immunodeficiency, infection of HIV, lymphoma, leukemia, SLE, JRA, inflammatory bowel disease or other autoimmune diseases.
* Received immunosuppressive therapy (such as long-term application of systemic glucocorticoids ≥ 14 days, dose ≥ 2 mg/kg/day or prednisone ≥ 20mg/day or equivalent to that dose of prednisone, excluding inhaled, intra-articular and topical steroid) within 3 months before vaccination.
* Serious cardiovascular diseases (pulmonary heart disease, pulmonary edema), liver and renal diseases and diabetes with complications.
* History of thrombocytopenia or other coagulation disorders, which may cause contraindications to intramuscular injection.
* Abnormal blood pressure (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) before vaccination; abnormal ECG
* Laboratory indicators out of the specified ranges (i.e., out of 1.5x of ULN or LLN), or with clinical significance as judged by the physician.
* Current/long-term history of alcohol abuse and/or history of drug abuse.
* Any other factors judged by investigator that may affect the safety of the subject or evaluation of the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of adverse reactions/events | 30 mins, 0-7 days, 8-30 days and 0-30 days
  Incidence rates of adverse reactions/events (ADRs/AEs)
Safety in terms of laboratory-based AEs | 3 days after each vaccination
  Incidence rates of abnormal laboratory indicators
Safety in terms of SAEs | Within 6 months after full vaccination
  Incidence rates of SAEs
Safety in terms of Adverse Events of Special Interest | Within 6 months after full vaccination
  Incidence rates of AESI

SECONDARY OUTCOMES:
Immunogencity in terms of GMT by ELISA or FAMA | Days 1, 30, 60, 90 and 240
  GMC of anti-gE antibody and GMT of anti-VZV antibody
Immunogencity in terms of Seroconversion Rates | Days 30, 60, 90 and 240
  Seroconversion rates of anti-gE and anti-VZV antibody responses
Immunogencity in terms of Geometric Mean Fold Increase | Days 30, 60, 90 and 240
  GMFI of anti-gE and anti-VZV antibody responses
Immunogencity in terms of Cellular immunity | Days 1, 90 and 240
  Frequency of CD4+ and CD8+T cells that express at least one cytokine